CLINICAL TRIAL: NCT03136874
Title: Motivations and Psychological Aspects of the Gametes' Donation
Acronym: DonDon
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 13 6860 07
Record Dates: First submitted 2017-03-03; First posted 2017-05-02 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Gametes Donors
Keywords: donors; gametes; motivation; psychological
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Donors who procreated
  Interventions: Other: Interview and questionaires
- Donors who don't procreated
  Interventions: Other: Interview and questionaires

INTERVENTIONS:
Other: Interview and questionaires — * Quantitative method : Two questionnaires will be used to define sociodemographic data, motivations and personality traits of donors.
  * Qualitative method : Clinical interviewing allows data collection adapted to study the motivations of sperm/egg donors, their representations, the experience and the inscription of the donation in their personal stories.

SUMMARY:
The main objective is to study donors' personality and motivations characteristics of the different recruitment methods and thus to answer questions related to the donation's approach, its representations as well as motivations and the profile of the donors.

DETAILED DESCRIPTION:
The methodology used is mixed with a quantitative and qualitative approach. The first one is a psychosocial approach with two groups: donors of gametes without children, and donors who have already procreated. Two questionnaires will be used in this survey. The first aims to study the donors' socio-personal characteristics and motivations. The latter studies donors' personality traits.

The second approach is qualitative by a clinical case study. It is a psycho-dynamic approach, taking into consideration the donor (men and women), with all their subjectivity, their personal and family history and their representations.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for gametes donation
* Less than 45 years for men
* Less than 37 years for women
* Affiliation to social service

Exclusion Criteria:

* Under guardianship, or trusteeship

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volonteers are recruted in the different CECOS. These subjects (who have already procreated, or not) are going to donate sperm/egg.
Sampling Method: Non-Probability Sample
Enrollment: 1002 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Assessment of motivations of candidates who have procreated and those who have not procreated. | 1 hour
  Assessed by collecting questionnaire data and comparison between both groups of candidates.

SECONDARY OUTCOMES:
Assessment of the psychological profile of donors. | 4 months
  Profile comparison between candidates who have procreated and those who have not.
Assessment of the psychological profile of the donors and their motivations. | 4 months
  Links between their psychological profile and their motivations.
Assessment of the possibility of gametes preservation and donation motivations. | 4 months
  To understand links between the possibility of gametes preservation and donation motivations.
Assessment of the ethical aspects of donation. | 4 months
  Links between and the ethical aspects of donation and whether or not they have procreated.
Assessment of the ethical aspects of donation and personality questionnaires. | 4 months
  Links between the ethical aspects of donation and personality questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Bujan, Pr, Principal Investigator — CECOS Hôpital Paule de Viguier
Locations (22):
- France (22):
  - CECOS Alsace Strasbourg, Schiltigheim, Alsace
  - CECOS Aquitaine Bordeaux, Bordeaux, Aquitaine
  - CECOS Rhône-Alpes Lyon, Lyon, Auvergne-Rhône-Alpes
  - CECOS Auvergne Clermont-Ferrand, Clermont-Ferrand, Auvergne
  - CECOS Basse-Normandie Caen, Caen, Basse-Normandie
  - CECOS Bretagne Rennes, Rennes, Brittany Region
  - CECOS Centre Tours, Tours, Centre-Val de Loire
  - CECOS Champagne-ardenne, Reims, Champagne-ardenne
  - CECOS Franche-Comté, Besançon, Franche-Comté
  - CECOS Franche-Comté, Dijon, Franche-Comté
  - CECOS Languedoc-Roussillon Montpellier, Montpellier, Languedoc-Roussillon
  - CECOS Lorraine Nancy, Nancy, Lorraine
  - CECOS Midi-Pyrénées Toulouse, Toulouse, Midi-Pyrénées
  - CECOS Nord Lille, Lille, Nord
  - CECOS Pays de la Loire Nantes, Nantes, Pays de la Loire Region
  - CECOS Picardie, Amiens, Picardie
  - CECOS Provence-Alpes-Côte d'Azur Marseille, Marseille, Provence-Alpes-Côte d'Azur Region
  - CECOS Provence-Alpes-Côte d'Azur, Nice, Provence-Alpes-Côte d'Azur Region
  - CECOS Rouen, Rouen, Seine-Maritime
  - CECOS Paris Jean Verdier, Bondy, Seine-Saint-Denis
  - CECOS Paris Cochin, Paris
  - CECOS Paris Tenon, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahuja KK, Mostyn BJ, Simons EG. Egg sharing and egg donation: attitudes of British egg donors and recipients. Hum Reprod. 1997 Dec;12(12):2845-52. doi: 10.1093/humrep/12.12.2845. PMID 9455866
- [Background] Cauvin P. [Motivations of oocytes donors]. Gynecol Obstet Fertil. 2009 Nov-Dec;37(11-12):934-41. doi: 10.1016/j.gyobfe.2009.09.003. Epub 2009 Oct 12. French. PMID 19819747
- [Background] Pennings G. Mirror gametes donation. J Psychosom Obstet Gynaecol. 2007 Dec;28(4):187-91. doi: 10.1080/01674820701656492. PMID 17966048
- [Background] Sydsjo G, Lampic C, Brandstrom S, Gudmundsson J, Karlstrom PO, Solensten NG, Thurin-Kjellberg A, Svanberg AS. Personality characteristics in a Swedish national sample of identifiable oocyte donors. BJOG. 2011 Aug;118(9):1067-72. doi: 10.1111/j.1471-0528.2011.02953.x. Epub 2011 Apr 11. PMID 21481152
- [Background] Sydsjo G, Lampic C, Brandstrom S, Gudmundsson J, Karlstrom PO, Solensten NG, Thurin-Kjellberg A, Skoog Svanberg A. Who becomes a sperm donor: personality characteristics in a national sample of identifiable donors. BJOG. 2012 Jan;119(1):33-9. doi: 10.1111/j.1471-0528.2011.03172.x. Epub 2011 Oct 18. PMID 22004406